CLINICAL TRIAL: NCT05990322
Title: Empowering Anxious Parents to Manage Child Avoidance Behaviors: A Randomized Trial of a Single-Session Intervention Targeting Parent Accommodation
Brief Title: Empowering Economically Insecure Parents to Manage Child Anxiety
Acronym: ProjectEmpower
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 00195
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Project EMPOWER; Online Resources and Referrals

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project EMPOWER (Experimental): Project EMPOWER is a web-based, self-administered SSI for parents that takes about 30 minutes to complete. The program includes 5 elements, based on current best-practices in SSI design (Schleider, Dobias, Sung, & Mullarkey, 2020) and existing interventions targeting accommodation (Lebowitz & Omer, 2014): (1) an introduction to the program's rationale; (2) psychoeducation around child anxiety and avoidance, along with how parental accommodation can inadvertently maintain child anxiety; (3) information on how parents can better identify children's patterns of avoidance and encourage brave behavior instead; (4) facilitating parents' creation of an "action plan" for promoting brave behavior and reduce avoidance in their own child; (5) a vignette exercise in which parents read about another family's difficulty managing their child's anxiety; parents identify the elements of the anxiety cycle and provide possible solutions to these parents based on what they learned.
  Interventions: Behavioral: Project EMPOWER
- Online Resources and Referrals (Placebo Comparator): Online Resources and Referrals (ORR) is an information sheet containing materials about the nature of child anxiety and a list of national resources related anxiety treatment. ORR does not include any psychoeducational components regarding parental accommodation.
  Interventions: Behavioral: Project EMPOWER

INTERVENTIONS:
Behavioral: Project EMPOWER — Experimental Condition

SUMMARY:
Efforts to develop and disseminate evidence based practices (EBPs) for youth anxiety have made great strides. Still, up to 82.2% of youth who need mental health treatment for anxiety never access care or drop out prematurely; commonly cited barriers to treatment are shortage of care, transportation limitations, financial burden, and gatekeeping behaviors by caretakers. As such, there is great need for accessible, scalable interventions that can ameliorate the global burden of youth anxiety, including those that help prevent the onset of anxiety in high-risk children. Single session interventions (SSIs), which have prevented and reduced child anxiety across numerous trials to date, may offer a promising solution, given their potential disseminability and cost-effectiveness. The proposed randomized trial will evaluate the effects of a novel, web-based, self-guided SSI designed to systematically reduce parent accommodation in economically insecure parents.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common, debilitating forms of childhood psychopathology, affecting 8.3-27.0% of youth before the age of 18 (Costello, Egger, & Angold, 2005). Child anxiety increases risk for psychiatric comorbidities across the lifespan (Copeland, Angold, Shanahan, & Costello, 2014), creates significant burdens for caregivers (Ramos-Cerqueira et al., 2008), and carries societal costs (Beecham, 2014; Bodden, Dirksen, Bögels, 2008). Although numerous interventions have been developed to treat youth anxiety disorders (Kendall, Achenbrand, & Hudson, 2003), up to 82.2% of US youth with anxiety will not receive adequate care (Merikangas et al., 2011). Several reasons may explain this discrepancy, including the length and cost of existing evidence-based interventions (EBIs) and limited accessibility for families in need. As such, there is great need for accessible, scalable interventions that can ameliorate the global burden of youth anxiety, including those that help prevent the onset of anxiety in high-risk children.

The inaccessibility of mental health care to low-SES children is especially problematic given the heightened risk for mental health problems within this population. (Bøe et al., 2011; Keating & Hertzman, 2000; Mendelson et al., 2008). In fact, children and adolescents who are socioeconomically disadvantaged are 3 times more likely to experience mental health difficulties, relative to their more advantaged peers (Reiss, 2013). This may reflect the fact that low SES is closely related to various other risk factors to psychopathology, like weaker family support networks, increased community violence exposure, greater odds of caregivers using harsh discipline strategies, and more exposure to stressful family life events (Everson-Rose et al., 2011; Hill et al., 1996; Shaw et al., 1998; Stein et al., 2003). Access levels vary as well; an examination of nation-wide data of mental health access among adolescents indicate that low-income families are significantly less likely to connect to services (Newacheck et al., 2003). Unfortunately, even when lower-SES youth do access evidence-based treatments, they may benefit less than their more-advantaged peers. It is critical to develop interventions that can not only efficiently target mechanisms most critical to reducing child psychopathology-especially common, impairing problems like anxiety disorders- that are designed for accessibility among historically underserved populations. A simultaneous emphasis on developing and testing child anxiety interventions that are effective and accessible is necessary to adequately serve the lower-SES children and families they are presumably designed to help.

Single-session interventions (SSIs) may offer one potential solution to this gap in care. SSIs include core components of comprehensive EBIs delivered succinctly to improve the odds of access and completion (Schleider & Weisz, 2017a). In a recent meta-analysis of 50 RCTs, SSIs reduced youth mental health problems of multiple disorders, with SSIs targeting child anxiety producing the largest effects (mean g = 0.58; Schleider & Weisz, 2017b). Thus, well-targeted SSIs may offer cost-effective additions or alternatives to traditional care for anxiety in youth. Given that family factors play a crucial role in the etiology of child anxiety, SSIs targeting parents and their interactions with offspring offer a novel approach to preventing youth anxiety (Degnan, Almas, Fox, 2010). Thus, the aim of this project is to test the acceptability and short-term effects of a novel, web-based SSI targeting parental accommodation: a well-established, potentially modifiable risk factor for child anxiety. Results may reveal a promising, targeted approach to scalable child anxiety prevention.

Research shows that parent accommodation can be systematically reduced via psychosocial intervention, and interventions targeting accommodation have helped mitigate child anxiety (Lebowitz, 2014). Translating core components of existing interventions that target parental accommodation into briefer, self-administered SSIs (i.e., those that do not involve a trained therapist) may improve families' access to empirically driven supports for child anxiety. It may also enhance the implementation of mental health interventions by lay providers who frequently interact with children (e.g. teachers and pediatricians). Thus, the goal of this project is to test a web-based, self-guided SSI (Project EMPOWER) targeting parental accommodation in a financially diverse sample.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one child between the ages of 4-10 years old
* Spouse/partner has not taken part of this study before
* Report clinical levels of child anxiety symptoms, per a score above a 7.5 on the Brief SPENCE Children's Anxiety Scale
* Report economic insecurity, indicated by a score less than or equal to 44 on the Consumer Financial Protection Bureau Financial Well-Being Scale (CFPB)

Exclusion Criteria:

* Participant is non-English speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Family Accommodation Scale | Change from Baseline to 2-week and 4-week follow up
  Family Accommodation Scale is a 9-item measure designed to assess the extent a caregiver accommodate a child's anxiety symptoms; example questions include: "how often did you assist your child in avoiding things that might make him/her more anxious?" and "have you modified your family routine because of your child's symptoms?" Items are rated from 0 (never) to 4 (daily). Scores range from 0-36 with higher scores indicating more frequent parental accommodation
Perceived pre-to-post SSI change | Immediately after the SSI
  This two-item measure assesses participants' perceived change in their ability to help their children manage distressing situations and their ability to provide validation to their children from pre- to post-SSI. Parents in both groups will rate this question on a 5-point scale of 1 (much less able) to 5 (much more able).

SECONDARY OUTCOMES:
Distress Tolerance Scale | Change from Baseline to 2-week and 4-week follow up
  16 item measure assessing the extent to which one experiences and withstand distressing emotional states. Each item is rated on a 5-point Likert scale from 1 (strongly agree) and 5 (strongly disagree). Total score ranges from 16 to 80 with a higher score indicating higher levels of distress tolerance.
Program Feedback Scale | Immediately after the SSI
  The program feedback scale asks participants to rate 7 statements regarding acceptability and feasibility; note whether they would recommend this activity to others; and share what they liked and would change about the SSI. The 7 statements are rated from 0 (Really Disagree) to 5 (Really Agree). Total score ranges from 0 to 35, with higher scores indicating a more positive program evaluation.
Penn State Worry Questionnaire | Baseline
  16 item self-report questionnaire that asks individuals to rate how typical worry-related problems are for them, from 1 (not at all typical) to 5 (very typical). Scores range from 16-80; higher scores indicate more severe worry.
Consumer Financial Protection Bureau Financial Well-Being Scale | Baseline
  The CFPB Financial Well-Being Scale measures financial well-being as it relates to control over finances, capacity to absorb financial shock, and having the financial freedom to enjoy life. Parents are asked to answer 10 questions on a 0 to 4 Likert scale to generate a sum score, which is converted into a standardized score. Scores range from 14 to 95 with higher scores indicating a higher level of measure financial well-being.
Brief SPENCE Children's Anxiety Scale | Change from baseline to 4-week follow-up
  8-item measure assessing the severity of child anxiety symptoms on 4 domains: generalized anxiety, separation anxiety, panic/agoraphobia, and social anxiety. Parents are asked to report on how often their child experiences each anxiety symptom on a scale of 0 (never) to 4 (always). Total score ranges from 0 to 32, with higher scores indicating higher levels of anxiety in each domain.
Strengths and Difficulties Scale | Baseline
  25-item questionnaire that ask parents to answer questions about their 4 to 17 year old child to screen for 5 domains: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior on a scale of 0 (not true) to 2 (certainly true). Total score ranges from 0 to 40 with higher scores indicating a higher severity of each domain
Parental Stress Scale | Baseline
  18 item measure of parental stress levels, parents rate on a scale of 1 (strongly disagree) to a 5 (strongly agree) scale on their perceived positive and negative experience of being a parent.
Everyday Discrimination Scale | Baseline
  5 item questionnaire used to assess subjective experiences of discrimination. Participants use a scale of 1 (never) to 5 (at least once a week) to rate how often they have experienced discrimination
Patient Health Questionnaire | Baseline
  Patient Health Questionnaire (PHQ-4) is a 4 item scale measuring anxiety and depression. Participants rate each statement on a scale of 0 (not at all) to 4 (nearly every day) to rate the severity of their worry and depression

IPD SHARING:
Plan to Share IPD: Undecided